CLINICAL TRIAL: NCT01680874
Title: A Pilot Study to Examine the Role of Probiotics for Improving Outcomes of C. Difficile
Brief Title: Probiotics for Clostridium Difficile Infection in Older Adults
Acronym: PICO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012-0462; R03AG040669-01 (NIH)
Record Dates: First submitted 2012-09-04; First posted 2012-09-07 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Clostridium Difficile
Keywords: Clostridium difficile; Diarrhea; Infection; Lactobacilli; Bifidobacteria; Lactobacillus acidophilus; Lactobacillus paracasei; Bifidobacterium lactis; Yogurt; Probiotics
MeSH Terms: conditions — Diarrhea; Infections | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Probiotic (Experimental): This arm will receive a probiotic combination which will consist of equal amounts of Lactobacillus acidophilus NCFM® (ATCC 700396), Lactobacillus paracasei Lpc-37 (ATCC SD5275), Bifidobacterium lactis Bi-07 (ATCC SC5220), and Bifidobacterium lactis Bl-04 (ATCC SD5219).
  The probiotic will be taken orally, once a week, for 4 weeks.
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): A placebo will be taken orally, once a day, for 4 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — The intervention will consist of the subject taking the study medication once a day for 4 weeks. During hospitalization, patients will be followed daily for diarrhea history, record of concomitant medications, adverse effects (AEs), and their response to treatment using a stool diary. Upon discharge from the hospital, patients will be contacted through weekly phone calls to assess diarrhea history, record of concomitant medications, adverse effects (AEs), and their response to treatment using a stool diary. At weeks 4 and 8, a stool sample will be collected, and the stool diary will be reviewed.
  Other Names: Lactobacillus acidophilus NCFM®; Lactobacillus paracasei Lpc-37; Bifidobacterium lactis Bi-07; Bifidobacterium lactis Bl-04; ATCC 700396; ATCC SD5275; ATCC SD5220; ATCC SD5219
  Arms: Probiotic
Dietary Supplement: Placebo — The intervention will consist of the subject taking the placebo once a day for 4 weeks. day for 4 weeks. During hospitalization, patients will be followed daily for diarrhea history, record of concomitant medications, adverse effects (AEs), and their response to treatment using a stool diary. Upon discharge from the hospital, patients will be contacted through weekly phone calls to assess diarrhea history, record of concomitant medications, adverse effects (AEs), and their response to treatment using a stool diary. At weeks 4 and 8, a stool sample will be collected, and the stool diary will be reviewed.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether a probiotic, when used together with standard treatment, is effective in reducing duration of symptoms and preventing recurrence of infection in older adults with a first episode of C. difficile infection.

DETAILED DESCRIPTION:
Probiotics are live microorganisms that are available over the counter, widely used as dietary supplements or nutritional foods, and represent a low-cost, well tolerated, safe, non-antibiotic based strategy that may have efficacy as adjunctive treatment of infections without the attendant risks of promoting antimicrobial resistance. Certain probiotics have demonstrated inhibition of adherence of pathogenic bacteria and stimulation of systemic immune functions, possibly enhancing the body's ability to eradicate C. difficile in the gastrointestinal tract. However, limited data is available on the efficacy of probiotics for ameliorating C. difficile symptoms and reducing recurrence of C. difficile infection (CDI). The investigators propose a pilot randomized, double-blind, placebo-controlled clinical trial in older adult inpatients with a first episode of CDI to evaluate the efficacy of a probiotic combination, in conjunction with standard treatment, for reducing duration of diarrhea and recurrence of CDI.

ELIGIBILITY:
Inclusion Criteria:

* Adult of either gender, 18 years or older with a first episode of C. difficile infection
* Meets the case definition of C. difficile infection-diarrhea associated with a positive stool test for C. difficile toxin(s) in the 2 days prior to enrollment treated with metronidazole or vancomycin

Exclusion Criteria:

* Severe disease defined as any of the following: WBC > 30,000 or < 1000 cells/mm^3, elevated creatinine > 1.5 times the premorbid level, ICU patient at time C. difficile infection diagnosed
* Has other known etiology of diarrhea (e.g. other enteric pathogen, other intestinal disease)
* Has a history of chronic intestinal disease (e.g. Crohn's disease, ulcerative colitis)
* Has a presence of toxic megacolon or ileus
* Has a presence of colostomy or nasogastric tube
* Has a history of abdominal surgery within the previous 3 months (from time of enrollment)
* Is enrolled in another investigational drug trial
* Is unavailable for follow-up visits
* History of multiple C. difficile infection
* Willing not to take other probiotics for duration of study
* Is severely immunocompromised.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-02; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Duration of diarrhea | 4 weeks
  Duration of diarrhea, as indicated by a stool diary kept by the patient

SECONDARY OUTCOMES:
Density of C. difficile toxin in stool | 8 weeks
Stool cytokines | 8 weeks
Fecal lactoferrin | 8 weeks
Functional assessment using Barthel Index | 8 weeks
Recurrence of CDI | 8 weeks
  Diagnosis with a recurrent episode of C. difficile infection

OTHER OUTCOMES:
Infection with Lactobacillus | 8 weeks
  Fever and other signs of infection with Lactobacillus, and infection confirmed through blood cultures
Infection with Bifidobacterium | 8 weeks
  Fever and other signs of infection with Bifidobacterium, and infection confirmed through blood cultures

CONTACTS AND LOCATIONS:
Overall Officials: Nasia Safdar, MD, Principal Investigator — University of Wisconsin Department of Medicine (Infectious Disease)
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

REFERENCES:
- [Background] Alvarez-Olmos MI, Oberhelman RA. Probiotic agents and infectious diseases: a modern perspective on a traditional therapy. Clin Infect Dis. 2001 Jun 1;32(11):1567-76. doi: 10.1086/320518. Epub 2001 May 4. PMID 11340528
- [Background] McFarland LV. Meta-analysis of probiotics for the prevention of antibiotic associated diarrhea and the treatment of Clostridium difficile disease. Am J Gastroenterol. 2006 Apr;101(4):812-22. doi: 10.1111/j.1572-0241.2006.00465.x. PMID 16635227
- [Background] Safdar N, Barigala R, Said A, McKinley L. Feasibility and tolerability of probiotics for prevention of antibiotic-associated diarrhoea in hospitalized US military veterans. J Clin Pharm Ther. 2008 Dec;33(6):663-8. doi: 10.1111/j.1365-2710.2008.00980.x. PMID 19138244
- [Derived] Barker AK, Duster M, Valentine S, Hess T, Archbald-Pannone L, Guerrant R, Safdar N. A randomized controlled trial of probiotics for Clostridium difficile infection in adults (PICO). J Antimicrob Chemother. 2017 Nov 1;72(11):3177-3180. doi: 10.1093/jac/dkx254. PMID 28961980
- [Derived] Barker A, Duster M, Valentine S, Archbald-Pannone L, Guerrant R, Safdar N. Probiotics for Clostridium difficile infection in adults (PICO): Study protocol for a double-blind, randomized controlled trial. Contemp Clin Trials. 2015 Sep;44:26-32. doi: 10.1016/j.cct.2015.07.015. Epub 2015 Jul 22. PMID 26210512